CLINICAL TRIAL: NCT02798380
Title: An Open-Label Phase 2 Study to Investigate the Efficacy, Tolerability, and Safety of the HTS-519 Insert in the Treatment of Subjects With Distal Lateral Subungual Onychomycosis of the Great Toenail
Brief Title: Efficacy, Safety, and Tolerability of HTS-519 Insert in Patients With Toenail Fungus of the Big Toenail
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hallux, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HTS-002B
Record Dates: First submitted 2016-06-05; First posted 2016-06-14 (Estimated); Results first posted 2019-09-24 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HTS-519 Insert (Experimental): Active treatment
  Interventions: Drug: HTS-519 Insert

INTERVENTIONS:
Drug: HTS-519 Insert — Maximum feasible dose of HTS-519 Insert per diseased nail
  Other Names: HTS-519 Biodegradable Micro Insert

SUMMARY:
The purpose of this study is to assess the efficacy, safety and tolerability of HTS-519 Inserts in the treatment of mild to moderate toenail fungus disease of the big toenail.

DETAILED DESCRIPTION:
Open label, single-site

ELIGIBILITY:
Inclusion Criteria:

* Male and females 18 - 74 years of age inclusive
* Fungal toenail infection of one or both of the large (great) toenails
* The nail infection must be due to a dermatophyte, (mixed infections [dermatophyte and non-dermatophyte] are not allowed)
* Willingness not to have professional pedicures or application of any nail polish product or nail cosmetics to the toenails after the screening visit

Exclusion Criteria:

* History of any significant chronic fungal disease other than onychomycosis or immunocompromised condition
* Any abnormalities of the nail or previous surgery of the toenail that could prevent a normal appearing nail if clearing of infection is achieved
* Significant confounding conditions as assessed by the study doctor
* Participation in any other trial of an investigational drug or device within 30 days or participation in a research study concurrent with this study
* No administration of systemic antifungal medications within 6 months prior to screening visit
* No application of prescription topical antifungal medications for toenail fungus within 3 months or other commercially available topical medications for toenail fungus applied directly to the toenails within 1 month prior to screening visit
* Tinea pedis (athlete's foot) that would require systemic treatment

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Tremblay, RN, BSN, Study Director — Hallux, Inc.
Locations (1):
- OrthoArizona - East Valley Foot & Ankle Specialists, Mesa, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HTS-519 Insert
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | HTS-519 Insert
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 12
Age, Continuous [Mean (Full Range); unit: years] | 59.9 [26 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Treatment Related Adverse Events
Description: Frequency and severity of Treatment Related Adverse Events
Time Frame: Up to 48 weeks
Population: Safety Population: All Enrolled
Measure: Count of Participants; unit: Participants
Groups:
- Safety Population: All Enrolled: Active treatment
  HTS-519 Insert: Maximum feasible dose of HTS-519 Insert per diseased nail
Arm/Group | Safety Population: All Enrolled
Number analyzed (Participants) | 30
Participants
  No. of Subjects with Treatment-related AE | 22
  No. of Subjects with no Treatment-related AE | 8

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | HTS-519 Insert
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 2/30
Other Adverse Events (participants affected / at risk) | 28/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HTS-519 Insert (N=30)
Leg edema (Investigations) | 1 (1) — Severe Right Leg Edema/ Not related
Spinal Fusion Surgery (Surgical and medical procedures) | 1 (1) — L4-S1 Spinal Fusion/ Not related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HTS-519 Insert (N=30)
Mild Punctate Bleeding (General disorders) | 4 — Preferred Term = Implant site haematoma
Mild Subungual Hematoma (General disorders) | 17 — Preferred Term = Implant site haemorrhage
Mild Pain in Toe (Investigations) | 2 — Preferred Term = Pain in Toe
Mild Onycholysis (Skin and subcutaneous tissue disorders) | 5 — Preferred Term = Onycholysis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-12): https://cdn.clinicaltrials.gov/large-docs/80/NCT02798380/Prot_SAP_001.pdf